CLINICAL TRIAL: NCT04145362
Title: Assessment of Factors Affecting Sleep-Wake Patterns in Preterm Infants by Actigraphy, Amplitude Integrated Electroencephalography (aEEG), Sleep Diaries and Direct Observation
Brief Title: Sleep-wake Patterns in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Perran Boran, Professor of Pediatrics, Marmara University
Other Study IDs: SAG-C-TUP-131217-0647
Record Dates: First submitted 2019-10-27; First posted 2019-10-30 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2019-10

CONDITIONS: Sleep
Keywords: preterm; actigraphy; sleep
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The development of sleep-wake behavior is considered to be one of the most important maturation processes occurring in the first year of life. Sleep-wake behavior is related to neurobehavioral regulation of the infant and cognitive function, and gives important information about infant's health. It is suggested that the identification of sleep-wake patterns in preterm infants is critical to the detection of future disorders, early diagnosis and planning of intervention studies In this study we aimed to recruit a total of 25 premature babies born between 28 to 37 weeks of gestational age over six month in the Neonatal Intensive Care Unit of Marmara University Pendik Training and Research Hospital. Sleep wake cycles of these premature infants will be assessed at 32 weeks corrected age by actigraphy, sleep diaries, direct observation and Amplitude integrated electroencephalography (aEEG). We also aimed to investigate the maturation of sleep patterns of these infants included in the study at postconceptional 40th weeks of age, and 12th, and at 24th weeks corrected age, by sleep diaries and actigraphic measurements at their home environment. Development will be assessed by Bayley and Ages and Stages Questionnaire.

DETAILED DESCRIPTION:
Studies show that the patterns of sleep-wakefulness reflect the maturation of the central nervous system in preterm infants and are indicative of behavioral development. It is emphasized that the identification of sleep-wake patterns in preterm infants is critical to the detection of future disorders, early diagnosis and planning of intervention studies.

The primary objective of this study is to assess factors affecting the maturation of sleep wake cycles in preterm infants by actigraphy, sleep diaries, direct observation, and aEEG. Our secondary objectives were to assess the neurodevelopment of these infants.

In this study we aimed to recruit a total of 25 premature babies born between 28 to 37 weeks of gestational age over a six month period in the Neonatal Intensive Care Unit of Marmara University Pendik Training and Research Hospital. Sleep architecture will be assessed at 32 corrected age by actigraphy, sleep diaries, and aEEG. Simultaneous video recording and direct observation will be performed and sleep stages will be defined. Anderson Behavioral State Scale will also be applied. Philips Respironics Actiwatch-2 devices will be used. The follow up will be at post conceptional 40 weeks, 12 and 24 weeks corrected age. Development will be assessed by Bayley test and Ages and Stages Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Being preterm admitted to Neonatal Intensive Care Unit
* Gestational age must be between 28 to 37 weeks

Exclusion Criteria:

* Preterm still receiving invasive mechanical ventilation at the time of data collection,
* Major congenital anomalies,
* Critically ill babies (sepsis),
* Major cerebral injuries (intraventricular hemorrhage grade III, and IV, periventricular leukomalacia)
* Retinopathy of prematurity grade III and IV,
* Necrotizing enterocolitis
* Infants using sedative or anticonvulsant drugs

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born between 28 to 37 weeks of gestational age
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Sleep architecture in preterm infants during their stay in Newborn Intensive Care Unit | 1 day of assessment
  Preterm infant's sleep wake patterns will be described by using actigraphy, aEEG, and video recorded direct observation
Preterm infant's sleep wake patterns will be described at 12, and 24 weeks of corrected age | 6 months corrected age
  Preterm infant's sleep wake patterns will be described at 12, and 24 weeks of corrected age by actigraphy, and sleep diaries

SECONDARY OUTCOMES:
Neurodevelopmental assessment using the Bayley Scales of Infant and Toddler development (Third Edition) | corrected age 6 months
  Bayley Scales of Infant and Toddler development (Third Edition) will be used for neurodevelopment assessment at 12, and 24 weeks of corrected age
Developmental screening using the Ages and Stages Questionnaire (ASQ-2) | corrected age 6 months
  Ages and Stages Questionnaire (ASQ-2) is parent-completed questionnaire that will be used as a general developmental screening tool

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ulgen O, Baris HE, Askan OO, Akdere SK, Ilgin C, Ozdemir H, Bekiroglu N, Gucuyener K, Ozek E, Boran P. Sleep assessment in preterm infants: Use of actigraphy and aEEG. Sleep Med. 2023 Jan;101:260-268. doi: 10.1016/j.sleep.2022.11.020. Epub 2022 Nov 20. PMID 36459917